CLINICAL TRIAL: NCT03230773
Title: Can Untrained Bystanders Safely and Effectively Use an Automated External Defibrillator (AED) in a Cardiac Arrest Scenario?
Brief Title: Use of Public Access Defibrillators by Untrained Bystanders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Postponed
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Charles D. Deakin, Professor of Resuscitation, University Hospital Southampton NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26783
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Arrest; Sudden Death, Cardiac
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Prospective, randomised study with volunteers randomised to use one of six different defibrillator designs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Defibrillator - Model 1 (Experimental): Time taken to open, attach and then discharge the defibrillator on a manikin during a simulated cardiac arrest scenario.
  Interventions: Device: Defibrillator model
- Defibrillator - Model 2 (Experimental): Time taken to open, attach and then discharge the defibrillator on a manikin during a simulated cardiac arrest scenario.
  Interventions: Device: Defibrillator model
- Defibrillator - Model 3 (Experimental): Time taken to open, attach and then discharge the defibrillator on a manikin during a simulated cardiac arrest scenario.
  Interventions: Device: Defibrillator model
- Defibrillator - Model 4 (Experimental): Time taken to open, attach and then discharge the defibrillator on a manikin during a simulated cardiac arrest scenario.
  Interventions: Device: Defibrillator model
- Defibrillator - Model 5 (Experimental): Time taken to open, attach and then discharge the defibrillator on a manikin during a simulated cardiac arrest scenario.
  Interventions: Device: Defibrillator model
- Defibrillator - Model 6 (Experimental): Time taken to open, attach and then discharge the defibrillator on a manikin during a simulated cardiac arrest scenario.
  Interventions: Device: Defibrillator model

INTERVENTIONS:
Device: Defibrillator model — Comparison of the performance of different public access defibrillators

SUMMARY:
Survival from out-of-hospital cardiac arrest is time critical and diminishes rapidly without appropriate intervention. Bystander CPR at least doubles the chances of survival and the additional use of a public access defibrillator (PAD) can again double overall survival rates. PADs are designed to be easy and simple to use, but whether untrained bystanders can use them safely and effectively is unknown. This study will aim to assess the ability of untrained bystanders to deploy a PAD in a simulated cardiac arrest.

DETAILED DESCRIPTION:
Survival from out-of-hospital cardiac arrest is time critical and diminishes rapidly without appropriate intervention. Overall survival is no more than 10% in the UK.

Bystander CPR at least doubles the chances of survival and the additional use of a public access defibrillator (PAD) can again double overall survival rates. Because PADs can make such a dramatic increase in chances of survival, public health programmes have encouraged the deployment of PADs in areas of high public density in order to deliver early defibrillation prior to ambulance arrival. Where this can be achieved, survival rates as high as 50% have been reported.

PADs are designed to be easy and simple to use, and in addition to graphical instructions on the device, give verbal instructions to a rescuer in order to ensure the PAD is used correctly. Most bystanders who are first on scene at a cardiac arrest have no first aid training and it is not always possible to wait for someone with first aid training to be available to use a PAD. Several guidelines, such as those from the Resuscitation Council (UK), state that untrained bystanders can use a PAD, but there has been little evaluation to understand whether this can safely and effectively be achieved without specific PAD training.

This study will aim to assess the ability of untrained bystanders to safely and effectively deploy a PAD in a simulated cardiac arrest, specifically aiming to identify differences between the features of different devices that improve their ease of use in order to understand what design features are required for optimal design.

ELIGIBILITY:
Inclusion Criteria:

* Members of the public who have never received any first aid (CPR) training

Exclusion Criteria:

* Those less than 16 yrs age
* Those with any physical disability precluding the use of a PAD

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Time from arrival at patient side to discharging a defibrillation shock | Within the 5 mins of the simulated cardiac arrest.
  Comparison of median time taken to achieve this endpoint for each type of defibrillator

SECONDARY OUTCOMES:
Time from arrival at patient side to correct application of self-adhesive defibrillation pads | Within the 5 mins of the simulated cardiac arrest.
  Comparison of median time taken to achieve this endpoint for each type of defibrillator
Following of written and verbal instructions to ensure safe use of device | Within the 5 mins of the simulated cardiac arrest.
  % rescuers using each type of defibrillator without causing risk to themselves (as judged by observer)